CLINICAL TRIAL: NCT06258304
Title: A Phase 1 Dose Escalation and Expansion Study of GIGA-564, a Minimally Blocking Anti-CTLA-4 Monoclonal Antibody, in Participants With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Dose Escalation and Expansion Study of GIGA-564 in Participants With Locally Advanced or Metastatic Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GigaGen, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GG-GIGA-564-001
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Advanced or Metastatic Solid Tumor Malignancies
Keywords: GIGA-564, CTLA-4
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GIGA-564: Dose Escalation (Phase 1A) (Experimental): Up to 5 dose levels [0.3, 1.0, 3.0, 10.0, and 20.0 milligrams per kilogram (mg/kg)] will be evaluated sequentially. Participants will receive GIGA-564 intravenously over at least 60 minutes on Day 1 of every 3 weeks (3 weeks = 1 cycle) for up to 4 cycles until time of confirmed disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
  Interventions: Drug: GIGA-564
- GIGA-564: Dose Expansion (Phase 1B) (Experimental): Dose expansion (Phase 1B) of selected dose levels may be initiated following the preliminary clearance of those specified dose levels from the dose escalation (Phase 1A) as determined by the Sponsor and SRC. Participants will receive up to 4 cycles of one of up to three tolerable dose levels of GIGA-564. GIGA-564 will be given intravenously over at least 60 minutes on Day 1 of every 3 weeks (3 weeks = 1 cycle) for up to 4 cycles until time of confirmed disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
  Interventions: Drug: GIGA-564

INTERVENTIONS:
Drug: GIGA-564 — Administered by intravenous infusion
  Arms: GIGA-564: Dose Escalation (Phase 1A)
Drug: GIGA-564 — Administered by intravenous infusion
  Arms: GIGA-564: Dose Expansion (Phase 1B)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of GIGA-564 and identify the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) level(s) of GIGA-564 in participants with metastatic or locally advanced solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent.
* Histologically or cytologically confirmed locally advanced or radiographically confirmed metastatic solid tumor malignancies ineligible for standard-of-care or refractory to or relapsing after at least one line of systemic therapy in the metastatic or advanced setting.
* Measurable disease on imaging as based on Response Evaluation Criteria in RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* Life expectancy greater than three months.
* Electrocardiogram (ECG) without evidence of clinically relevant abnormalities in rhythm, conduction, or morphology of resting ECG or active ischemia as determined by the Investigator.
* Acceptable organ and marrow function including:

  1. Absolute neutrophil count >= 1,500 cells/ microliters (μL)
  2. Platelets >= 100,000 cells/μL
  3. Hemoglobin >= 9 grams per decilitre (g/dL)
  4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (≤ 3 × ULN if attributable to known Gilbert's syndrome)
  5. Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5 × ULN. If liver metastasis is present, AST/ALT < 5 × ULN
  6. Measured creatinine clearance ≥ 30 milliliter per minute mL/min per Cockcroft-Gault formula
  7. Prothrombin time or international normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1.5 × ULN, unless receiving anti-coagulant therapy.
* Primary or metastatic lesions that are amenable to biopsy (Phase 1B only).
* Women of childbearing potential must agree to use highly effective contraception.

Exclusion Criteria:

* Investigational therapy and/or anti-cancer therapy with the potential for late onset toxicity within 4 weeks or 5 half-lives (whichever is shorter), or nitrosoureas or mitomycin C within 6 weeks. Food and drug administration (FDA)-approved hormonal therapies (e.g., androgen deprivation therapy [ADT] for prostate cancer, anti-estrogen for breast cancer, somatostatin analogue for neuroendocrine cancer) are allowed.
* Failure to resolve toxicity from previous anti-cancer therapy (other than National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v5.0 ≤ Grade 2 alopecia, neuropathy or medically controlled endocrinopathies) to NCI CTCAE v5.0 ≤ Grade 1.
* Prior receipt of therapy directed against CTLA-4.
* Prior receipt of therapy directed against chemokine (C-C motif) receptor 8 (CCR8), cluster of differentiation 25 (CD25), or T cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine-based inhibition motif domains (TIGIT) with an active Fc domain.
* Baseline prolongation of corrected QT interval (QTc) QT/QTc interval Fridericia's formula (QTcF > 470 millisecond [msec]).
* History of hepatitis B (HBV) infection unless viral load is undetectable.
* Participants with known history of hepatitis C (HCV) infection, unless they have been treated and cured (viral load is undetectable).
* Active or severe infection such as active tuberculosis.
* Human immunodeficiency virus (HIV) infection unless participants are stable on anti-retroviral therapy (CD4 count ≥ 200/μL) and have a viral load < 400 copies/mL.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater heart failure), myocardial infarction within 3 months prior to initiation of study treatment, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Active or history of autoimmune or primary immunodeficiency disease requiring systemic treatment within 2 years of commencing study (NOTE: participants with autoimmune conditions requiring hormone replacement therapy or topical treatments are eligible).
* Active or history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of hematopoietic stem cell transplantation (HSCT) or solid organ transplant with the exception of corneal transplants.
* Pregnant or breastfeeding.
* Previous hypersensitivity reactions to any component of the investigational product.
* Concurrent use of systemic steroids (within 10 days of enrollment), except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids (e.g., in participants with exacerbations of reactive airway disease) must have completed therapy ≥ 10 days prior to enrollment. Steroid use to prevent intravenous contrast allergic reaction or anaphylaxis in participants who have known contrast allergies is allowed at any time prior to enrollment and for imaging while on treatment.
* History of other active malignancy within 3 years of enrollment except for the following: adequately treated localized skin cancer, ductal carcinoma in situ, cervical carcinoma in situ, superficial bladder cancer or other localized malignancy which has been adequately treated.
* Active or untreated brain metastases that are not stable. Stable is defined as 2 brain images that show no progression, obtained ≥ 4 weeks apart and any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved. Any steroids administered as part of this therapy must be completed ≥ 10 days prior to first dose of study medication.
* Thymoma or thymic carcinoma (Phase 1A only).
* Other medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and which, in the judgment of the Investigator or Sponsor, would make the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to 154 days
Number of Participants With Grade 3 or 4 TEAEs | Up to 154 days
Number of Participants With Treatment-related TEAEs | Up to 154 days
Number of Participants With Grade 3 or 4 Treatment-related TEAEs | Up to 154 days
Number of Participants With Serious Adverse Events (SAE's) | Up to 154 days
Number of Participants Who Discontinued Treatment due to Adverse Events (AEs) | Up to 154 days
Number of Participants With Dose-limiting Toxicities (DLTs) during Cycle 1 | Up to 21 days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to Week 24
Percentage of Participants with Minor RECIST 1.1 Response | Up to Week 24
Disease Control Rate (DCR) per RECIST 1.1 | Up to Week 24
Progression Free Survival (PFS) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Area Under the Serum Concentration-time Curve during a Dosage Interval (AUC0-tau) of GIGA-564 during Cycle 1 and Cycle 4 | Up to 84 days
Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC[0-inf)] of GIGA-564 during Cycle 1 | Up to 21 days
Maximum Observed Serum concentration (Cmax) of GIGA-564 during Cycle 1 and Cycle 4 | Up to 154 days
Time to Reach Maximum Observed Serum Concentration (Tmax) of GIGA-564 during Cycle 1 and Cycle 4 | Up to 154 days
Trough Observed Serum Concentration (C trough) of GIGA-564 during Cycle 1 and Cycle 4 | Up to 154 days
Elimination Half-life (t1/2) of GIGA-564 during Cycle 1 and Cycle 4 | Up to 154 days
Apparent Total Body Clearance (CL) of GIGA-564 during Cycle 1 | Up to 21 days
Volume of Distribution at Steady State (Vss) of GIGA-564 during Cycle 1 | Up to 21 days
Accumulation Ratio for Maximum Observed Serum Concentration (Cmax) of GIGA-564 | Up to 154 days
Accumulation Ratio for Trough Observed Serum Concentration (Ctrough) of GIGA-564 | Up to 154 days
Accumulation Ratio for Area Under the Serum Concentration-time Curve (AUC) of GIGA-564 | Up to 154 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No